CLINICAL TRIAL: NCT06977724
Title: A Phase1b, Multiple Ascending Dose, Open-label, Non-randomized Study Evaluating the Pharmacokinetics, Safety, and Efficacy of ABBV-319 in Subjects With Systemic Lupus Erythematosus (SLE) and Sjogren's Disease (SjD)
Brief Title: A Study to Assess Adverse Events, How the Drug Moves Through the Body and Effectiveness of Intravenous Infusions of ABBV-319 in Adult Participants With Systemic Lupus Erythematosus (SLE) and Sjogren's Disease (SjD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M25-433; 2024-519157-10 (Other: EU CT)
Record Dates: First submitted 2025-05-12; First posted 2025-05-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dry Eye Syndrome; Systemic Lupus Erythematosus
Keywords: Dry Eye Syndrome; Systemic Lupus Erythematosus; ABBV-319
MeSH Terms: conditions — Dry Eye Syndromes; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- ABBV-319 Group 1: SLE Participants (Experimental): Systemic Lupus Erythematosus (SLE) participants will receive 2 doses of ABBV-319 Dose A 21 days apart.
  Interventions: Drug: ABBV-319
- ABBV-319 Group 2: SLE Participants (Experimental): SLE participants will receive 2 doses of ABBV-319 Dose B 21 days apart.
  Interventions: Drug: ABBV-319
- ABBV-319 Group 3: SLE Participants (Experimental): SLE participants will receive 2 doses of ABBV-319 Dose C 21 days apart.
  Interventions: Drug: ABBV-319
- ABBV-319 Group 4: SLE Participants (Experimental): SLE participants will receive 2 doses of ABBV-319 Dose D 21 days apart.
  Interventions: Drug: ABBV-319
- ABBV-319 Group 5: SjD Participants (Experimental): Sjogren's disease (SjD) participants will receive 2 doses of ABBV-319 Dose TBD 21 days apart.
  Interventions: Drug: ABBV-319
- ABBV-319 Group 6: SjD Participants (Experimental): SjD participants will receive 2 doses of ABBV-319 Dose TBD 21 days apart.
  Interventions: Drug: ABBV-319

INTERVENTIONS:
Drug: ABBV-319 — Intravenous (IV) Infusion

SUMMARY:
Systemic lupus erythematosus (SLE) is a chronic, systemic autoimmune disease characterized by B cell hyperactivity and Sjorgren's disease (SjD) is a chronic, multisystem autoimmune disease characterized by lacrimal and salivary gland inflammation, with resultant dryness of the eyes and mouth and occasional glandular enlargement. ABBV-319 exhibits potential B cell depletion in SLE and SjD which are characterized by B cell hyperactivity. The purpose of this study is to assess the pharmacokinetics, safety, and efficacy of ABBV-319 in adult participants with SLE or SjD.

ABBV-319 is an investigational drug being developed for the treatment of SLE and SjD. Participants are placed in 1 of 6 groups called treatment arms. Each group receives a different dose of ABBV-319 depending on whether they have SLE or SjD. Around 36 adult participants with SLE or SjD will be enrolled at approximately 10 sites worldwide.

Participants will receive 2 doses of IV ABBV-319 21 days apart and will be followed for up to 343 days.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Lupus Erythematosus (SLE) Population - Clinical diagnosis of SLE at least 6 months prior to Screening as defined by the 2019 European Alliance of Associations for Rheumatology (EULAR)/American College Of Rheumatology (ACR) classification criteria for SLE and a positive antinuclear antibody (ANA) >= 1:80 drawn at Screening.
* SLE Population - Presence of anti-double stranded DNA (dsDNA), anti-Smith (Sm), anti-ribonucleoprotein (RNP), or anti-Sjogren's syndrome Ag A (SSA) Abs above the upper limit of normal (ULN).
* Sjogren's Disease (SjD) Population - Primary diagnosis of SjD at least 6 months prior to Screening as defined by the ACR/EULAR 2016 Criteria.
* SjD Population - EULAR Sjogren's Syndrome Disease Activity Index (ESSDAI) >= 5 at Screening.
* SjD Population - EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) >= 5 at Screening.

Exclusion Criteria:

* History of infection as defined in the protocol.
* Any of the medical diseases or disorders listed in the protocol.
* History of clinically significant (per investigator's judgment) drug or alcohol abuse within the 6 months prior to Screening.
* Any planned elective surgery that would impact study procedures or assessments through the completion of the Day 365 assessments.
* Any clinically significant ECG abnormalities at Screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to approximately 400 days
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.
Change from Baseline in B Cells in Blood and Tissue | Up to approximately 400 days
  Change from baseline in B cells in blood and tissue.
Maximum Plasma Concentration (Cmax) of ABBV-319 | Up to approximately 400 days
  Cmax of ABBV-319.
Time to Cmax (Tmax) of ABBV-319 | Up to approximately 400 days
  Tmax of ABBV-319.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-319 | Up to approximately 400 days
  t1/2 of ABBV-319.
Area Under the Concentration-Time Curve From Time 0 to Last Measurable Concentration (AUCt) of ABBV-319 | Up to approximately 400 days
  AUCt of ABBV-319.
Percentage of Participants with Detection of Anti-Drug Antibodies (ADAs) for ABBV-319 | Up to approximately 400 days
  Percentage of participants with detection of ADAs for ABBV-319.
Percentage of Participants with Detection of Neutralizing Antibodies (nAbs) for ABBV-319 | Up to approximately 400 days
  Percentage of participants with detection of nAbs for ABBV-319.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (4):
- United States (3):
  - Life Clinical Trials /ID# 276050, Margate, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 275836, Tampa, Florida
  - Private Practice - Dr. Ramesh C. Gupta I /ID# 275826, Memphis, Tennessee
- Amsterdam UMC, locatie AMC /ID# 274286, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-433